CLINICAL TRIAL: NCT03254862
Title: Investigation of Different Stimulation Patterns to Reduce Muscle Fatigue During Functional Electrical Stimulation (FES)
Brief Title: Different Stimulation Patterns to Reduce Muscle Fatigue During FES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Initial difficulties recruiting + main researcher had to withdraw from the study
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GN17NE114
Record Dates: First submitted 2017-08-16; First posted 2017-08-21 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Spinal Cord Injuries
Keywords: Functional electrical stimulation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: CSS & AsynS (Experimental): Electrical stimulation training on both legs:
  Conventional synchronous stimulation (CSS) and Asynchronous Sequential Stimulation (ASynS) - CSS/ASynS
  Interventions: Procedure: CSS/AsynS
- Group B: CSS & AsynR (Experimental): Electrical stimulation training on both legs:
  Conventional synchronous stimulation (CSS) and Asynchronous Random Stimulation (ASynR) - CSS/ASynR
  Interventions: Procedure: CSS/AsynR

INTERVENTIONS:
Procedure: CSS/AsynS — 16 sessions of training over a 4 week period consisting of repeated intermittent electrical stimulation (300ms On and 700ms Off stimulation) for 10 - 30 minutes. Conventional synchronous stimulation (CSS) on one leg; Asynchronous Sequential Stimulation (ASynS) on the other leg
  Arms: Group A: CSS & AsynS
Procedure: CSS/AsynR — 16 sessions of training over a 4 week period consisting of repeated intermittent electrical stimulation (300ms On and 700ms Off stimulation) for 10 - 30 minutes. Conventional synchronous stimulation (CSS) on one leg; Asynchronous Random Stimulation (ASynR) on the other leg.
  Arms: Group B: CSS & AsynR

SUMMARY:
The main aim of this study is to investigate the effect of patterned distribution stimulation compared to conventional stimulation in reducing muscle fatigue during functional electrical stimulation (FES) following spinal cord injury (SCI).

DETAILED DESCRIPTION:
Functional electrical stimulation (FES) is a commonly used technique in rehabilitation and often associated with rapid muscle fatigue which becomes the limiting factor in its applications. The main objective of this study is to investigate the effects on the onset of fatigue of conventional synchronous stimulation, as well as asynchronous stimulation that mimic voluntary muscle activation targeting different motor units which are activated sequentially or randomly via multiple pairs of stimulation electrodes. Three different approaches with various electrode configurations will be investigated, as well as different patterns of stimulation applied to the gastrocnemius muscle. In addition, the muscle changes during different patterns of stimulation will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* incomplete spinal cord injury
* able to give informed consent
* able to sit up in a chair

Exclusion Criteria:

* female subjects who are pregnant
* significant history of autonomic dysreflexia
* unable to give informed consent
* individuals who have a cardiac history
* individuals who have significant cognitive impairment
* individuals with muscular abnormality
* individuals who have significant contractures in the lower extremities
* individuals who have a rash or infection at the site of electrode placement (gastrocnemius for both legs)
* individuals who are hypersensitive to electrical stimulation
* individuals who are presently involved in another study which has overlap with the methodology and/or outcomes of the studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Muscle contraction ability | Baseline to 6 weeks
  Change in torque produced during muscle contraction

SECONDARY OUTCOMES:
Normalized Fatigue Index (NFI) | Baseline to 6 weeks
  Change in score on Normalized Fatigue Index (NFI)
Fatigue Time Interval (FTI) | Baseline to 6 weeks
  Change in Fatigue Time Interval (FTI)
Twitch-Tetanus Ratio response (ΔTTR) | Baseline to 6 weeks
  Change in Twitch-Tetanus Ratio response (ΔTTR)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Gollee, DipIng PhD, Study Director — University of Glasgow
Locations (1):
- Queen Elizabeth National Spinal Injuries Unit, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No